CLINICAL TRIAL: NCT01519271
Title: A Phase IV Randomized, Double-Blind, Placebo-Controlled, Crossover Single Site Study Of Exelon® Patch (Rivastigmine Transdermal System) For Mild Cognitive Impairment In Parkinson's Disease
Brief Title: Mild Cognitive Impairment in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 813803
Record Dates: First submitted 2012-01-10; First posted 2012-01-26 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: Parkinson's Disease; Mild Cognitive Impairment; Cognition; Memory; Attention; Exelon; Rivastigmine
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Patch (Placebo Comparator)
  Interventions: Drug: Placebo Patches
- Exelon Patch (rivastigmine transdermal system) (Active Comparator)
  Interventions: Drug: Exelon Patch (rivastigmine transdermal system)

INTERVENTIONS:
Drug: Exelon Patch (rivastigmine transdermal system) — The Exelon Patch (rivastigmine transdermal system) is a Cholinesterase Inhibitor approved by the FDA to treat Alzheimer's and Parkinson's Disease Dementia.
  5-10cm2 (4.6-9.5 mg of rivastigmine/24 hours )
  Arms: Exelon Patch (rivastigmine transdermal system)
Drug: Placebo Patches — The placebo patches will appear identical to the medication patches however they will be inactive (they will not contain rivastigmine).
  Arms: Placebo Patch

SUMMARY:
Mild cognitive impairment, including difficulty with solving problems, planning, attention, or recalling information, can be a significant problem for individuals with Parkinson's disease. Even mild cognitive difficulties can lead to worse functioning, quality of life, depression, and difficulty for caregivers. Thus, ideally treatment at this stage would improve both cognitive symptoms and some of the other problems associated with these symptoms.

Despite the fact that mild cognitive impairment is a serious problem for Parkinson's disease patients little is known about how best to treat it. This study is a 24-week clinical trial to see if a Food and Drug Administration (FDA)-approved drug, the Exelon (rivastigmine) Patch, is useful in treating mild cognitive impairment in patients with Parkinson's disease. Currently, the Exelon (rivastigmine) Patch is FDA-approved for the treatment of mild to moderate dementia in Alzheimer and Parkinson's disease patients.

DETAILED DESCRIPTION:
This study has 2 phases. Each phase will last 10 weeks and there will be a 4-week break between the 2 phases. Thus, you will be enrolled in the study for a total of 24 weeks. Over the course of the 24-week period we will schedule to see you in-person 6 times and check-in with you on the telephone 4 times, 2 times during each phase.

Phase I

Screening (may be the same day as the baseline visit) - Research personnel will determine if you are eligible to participate in this study.

Visit 1 - Baseline Visit, Start Study Medication

Phone Call 1 - Check in to see how you are feeling after starting the study medication

Visit 2 - 4 Weeks after Baseline, Increase Study Medication if tolerated

Phone Call 2 - Check in to see how you are feeling after increasing the study medication

Visit 3/ Phase I Termination Visit - 10 Weeks after Baseline (Phase I Termination Visit)

4 Week Break (no study medication)

Phase II

Visit 4/ Phase II Baseline - 14 Weeks after Baseline, Start Study Medication

Phone Call 3 - Check in to see how you are feeling after starting the study medication

Visit 5 - 18 Weeks after Baseline, Increase Study Medication

Phone Call 4 - Check in to see how you are feeling after increasing the study medication

Visit 6/Phase II and Study Termination Visit - 24 Weeks after Baseline

Visits 1, 3, 4, and 6 will last for about 2 ½ hours and visits 2 and 5 about 30 minutes. The 'check in' phone calls will last approximately 5-10 minutes.

After 24 weeks, your study participation will be over.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be experiencing symptoms of mild cognitive impairment; this will be determined by study personnel.
2. Participants must be on a sable medication regimen for 2 months prior to starting the study (necessary dose adjustments during the study are acceptable).
3. Participants are capable of giving informed consent supported by not meeting Parkinson's disease Dementia criteria; this will be determined by study personnel.

Exclusion Criteria:

1. Active suicide ideation.
2. Weighing less than 100 lbs (45 kgs).
3. History of Deep Brain Stimulation surgery.
4. Diagnosis of Dementia
5. Taking certain types of medications may be an exclusion criteria, this will be reviewed with all potential participants.
6. Females that are pregnant, planning to become pregnant, or are breastfeeding will not be included in the study. Females of childbearing potential will need to verify that they are not pregnant by a negative urine pregnancy test.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weintraub, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Ralston House, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Published Study Abstract — https://www.ncbi.nlm.nih.gov/pubmed/25914281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were a convenience sample of PD patients primarily from the Parkinson's Disease and Movement Disorders Center at the University of Pennsylvania. Patients between the ages of 40 and 85 y with idiopathic PD for more than 2 years and reporting cognitive were screened for study participation.
Pre-assignment Details: 48 participants assessed for eligibility, 28 randomized (17 did not meet inclusion/exclusion criteria and 3 refused to participate after screening)
Groups:
- Placebo First Then Rivastigmine: Placebo patches placed on skin daily in Phase 1 and Rivastigmine 5-10cm2 patches in Phase 2. Each phase lasted for 10 weeks.
  Exelon Patch (rivastigmine transdermal system): The Exelon Patch (rivastigmine transdermal system) is a Cholinesterase Inhibitor approved by the FDA to treat Alzheimer's and Parkinson's Disease Dementia.
  5-10cm2 (4.6-9.5 mg of rivastigmine/24 hours )
  Placebo Patches: The placebo patches will appear identical to the medication patches however they will be inactive (they will not contain rivastigmine).
- Rivastigmine First Then Placebo: 5-10cm2 rivastigmine patch daily first in phase 1 and placebo patch daily in phase 2. Each phase lasted for 10 weeks.
  Exelon Patch (rivastigmine transdermal system): The Exelon Patch (rivastigmine transdermal system) is a Cholinesterase Inhibitor approved by the FDA to treat Alzheimer's and Parkinson's Disease Dementia.
  5-10cm2 (4.6-9.5 mg of rivastigmine/24 hours )
  Placebo Patches: The placebo patches will appear identical to the medication patches however they will be inactive (they will not contain rivastigmine).
Period: Phase 1
Arm/Group | Placebo First Then Rivastigmine | Rivastigmine First Then Placebo
Started | 14 | 14
Completed | 14 | 13 (1 participant discontinued participation in the middle of phase 1.)
Not Completed | 0 | 1
Period: Phase 2
Arm/Group | Placebo First Then Rivastigmine | Rivastigmine First Then Placebo
Started | 12 (2 participants discontinued after Phase 1) | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Patch First Then 5-10cm2 Rivastigmine Patch: Placebo Patches: The placebo patches will appear identical to the medication patches however they will be inactive (they will not contain rivastigmine).
  Exelon Patch (rivastigmine transdermal system): The Exelon Patch (rivastigmine transdermal system) is a Cholinesterase Inhibitor approved by the FDA to treat Alzheimer's and Parkinson's Disease Dementia.
  5-10cm2 (4.6-9.5 mg of rivastigmine/24 hours )
  Each phase lasted 10 weeks.
- 5-10cm2 Rivastigmine Patch First First Then Placebo Patch: Exelon Patch (rivastigmine transdermal system): The Exelon Patch (rivastigmine transdermal system) is a Cholinesterase Inhibitor approved by the FDA to treat Alzheimer's and Parkinson's Disease Dementia.
  5-10cm2 (4.6-9.5 mg of rivastigmine/24 hours )
  Placebo Patches: The placebo patches will appear identical to the medication patches however they will be inactive (they will not contain rivastigmine).
  Each phase lasted 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Patch First Then 5-10cm2 Rivastigmine Patch | 5-10cm2 Rivastigmine Patch First First Then Placebo Patch | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (5.5) | 62.6 (10.1) | 64.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Cooperative Study- Clinical Global Impression Change (ADCS-CGIC)
Description: The ADCS-CGIC is the most commonly used measure of global change in dementia psychopharmacology studies. This assessment is a measure of change, thus it is not appropriate for baseline administration and only administered at the end of phase visit.
  The scale rates total improvement on a 7 point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
  A participant scoring a 1 or 2 is considered a responder on the CGI scale.
Time Frame: The ADCS-CGIC will be administered at the end of each study phase.
Population: Please note this study utilized the crossover design (i.e. participants were exposed to two phases of treatment, one with placebo and one with Exelon patch). The data are comparing differences in treatment groups. Over the course of this study 2 participants discontinued study participation.
Measure: Mean (Standard Deviation); unit: scores on the CGIC
Arm/Group | Placebo Patch | Exelon Patch (Rivastigmine Transdermal System)
Number analyzed (Participants) | 26 | 28
scores on the CGIC | 3.92 (0.94) | 3.48 (0.89)

2. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The MoCA will be used as the global cognitive screening instrument. It will also be administered in the clinical trial at baseline and the final visits of each phase as a secondary outcome measure of global cognition. Scores on the MoCA range from 0-30 with 26-30 indicating normal global cognition.
Time Frame: The MoCA was administered in the beginning and end of each study phase.
Population: Please note this study utilized the crossover design (i.e. participants were exposed to two phases of treatment, one with placebo and one with Exelon patch). The data are comparing differences in treatment groups.
Measure: Mean (Standard Deviation); unit: Score on MoCA
Groups:
- Placebo: Placebo Patches: The placebo patches will appear identical to the medication patches however they will be inactive (they will not contain rivastigmine).
- Rivastigmine: Exelon Patch (rivastigmine transdermal system): The Exelon Patch (rivastigmine transdermal system) is a Cholinesterase Inhibitor approved by the FDA to treat Alzheimer's and Parkinson's Disease Dementia.
  5-10cm2 (4.6-9.5 mg of rivastigmine/24 hours )
Arm/Group | Placebo | Rivastigmine
Number analyzed (Participants) | 23 | 23
Score on MoCA
  Baseline | 25.08 (2.7) | 24.93 (2.5)
  Week 16 | 24.73 (3.7) | 25.6 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Rivastigmine; Test type: Superiority; Cohen's D = .35

ADVERSE EVENTS:
Time Frame: Adverse events were recorded at every study visit post baseline (Phase 1: Week 4 and Week 10; Phase 2: Week 14, Week 18 and Week 24).
Description: We used a modified version of the Treatment Emergent Symptom Scale (TESS) to assess psychiatric, cognitive, and motor adverse effects.
Arm/Group | Placebo Patch | Exelon Patch (Rivastigmine Transdermal System)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 9/26 | 11/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Patch (N=26) | Exelon Patch (Rivastigmine Transdermal System) (N=28)
Increased Blood Pressure (Vascular disorders) | 6 | 8
Pain (General disorders) | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Other (General disorders) | 9 | 11
Tremor (Nervous system disorders) | 3 | 5
Decreased Blood Pressure (Vascular disorders) | 3 | 4
Fatigue (General disorders) | 2 | 4
Insomnia (General disorders) | 2 | 4
Worse Balance (Nervous system disorders) | 4 | 4
Visual Hallucinations (Psychiatric disorders) | 2 | 3
Increased "off" time (Nervous system disorders) | 1 | 3
Weight Loss (General disorders) | 3 | 1
Cognitive Impairment (General disorders) | 3 | 0
Depression (General disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
The small sample size may have limited our power to detect a treatment effect.

When the study was conducted, the maximum strength of the rivastigmine patch was 9.5 mg/24 h. Since then, a higher dose has been approved by the FDA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No